CLINICAL TRIAL: NCT05711303
Title: A Randomised, Double-blinded, Parallel, Placebo-controlled Study to Investigate the Effect of Superba Boost (Krill Oil Concentrate) on Various Skin Parameters in Healthy Adult Subjects
Brief Title: Study to Investigate the Effect of Superba Boost on the Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: AFCRO-097
Record Dates: First submitted 2019-06-25; First posted 2023-02-03 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Trans-epidermal Water Loss

STUDY DESIGN:
Intervention Model Description: Subjects who successfully meet the eligibility criteria will be randomized on a 1:1 basis, to receive Superba Boost or Placebo.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Randomization will be carried out by computer-generated block-randomization lists. Subjects will be randomized to one of the two treatment groups, in blocks of 6. The randomization will be seeded, with the seed only available to the statistician generating the randomization list.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superba Boost (Active Comparator): One 1000 mg capsule per day Superba Boost for 12 weeks
  Interventions: Dietary Supplement: Superba Boost
- Placebo (Placebo Comparator): One 1000 mg capsule per day placebo for 12 weeks
  Interventions: Dietary Supplement: Superba Boost

INTERVENTIONS:
Dietary Supplement: Superba Boost — To assess changes in Trans-epidermal water loss (TEWL), measured at baseline and after 12 weeks of intervention using a TEWAMetre.
  Other Names: Placebo

SUMMARY:
Study to determine the effect of 12 weeks daily consumption of Superba Boost as compared to placebo on reduction in Trans-Epidermal Water-Loss (TEWL).

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, parallel group trial in 70 healthy adult male and female subjects between 20 and 50 years. The primary objective is to assess whether Superba Boost krill oil administered at a dose of 1 g per day for 12 weeks (84 days) has a positive effect on the TEWL, skin hydration and elasticity. At screening, the subjects must have TEWL values of >10 g/m2/h and <24.9 g/m2/h when measured by a TWEAmeter, i.e. within the range defined as normal and healthy skin. The change in omega-3 index, defined as EPA and DHA as percentage of total fatty acids in red blood cells, will be measured and correlated to the changes in the skin parameters. The study consists of 4 visits: the screening visit (V1), baseline visit / week 0 / Start of treatment (V2), Interim / Week 6 (V3) and week 12 / end of treatment (V4) . In this study, subjects must have a low habitual consumption of fatty fish and seafood, defined as a frequency of twice per month or less will be recruited.

Each subject must fulfill all inclusion criteria and will not be allowed to meet any of the exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion, the subject must fulfil all of the following criteria:

1. Be able to give written informed consent;
2. Be aged between 20 and 50 years, inclusive;
3. Trans-epidermal water loss score >10 and ≤ 24.9 g/m²/h;
4. Be in general good health with no existing co-morbidities
5. Have a low habitual consumption of fatty fish and seafood, defined as a frequency of twice per month or less;
6. Be willing to avoid all fish and seafood meals in the 4-days before each scheduled clinic visit;
7. Be willing to maintain dietary habits and physical activity levels throughout the trial period;
8. Be able to communicate well with the Investigator, to understand and comply with the requirements of the study, and be judged suitable for the study in the opinion of the Investigator;
9. Willing & able to consume the investigational product daily for the duration of the study.

Exclusion Criteria:

The presence of any of the following criteria will exclude the subject from participating in the study:

1. Pregnant or breastfeeding women; women planning to become pregnant during the study;
2. Women of child-bearing potential who do not use an acceptable method of contraception;
3. Suffer from photosensitivity;
4. History of skin cancer;
5. Are currently taking photosensitizing medication, or have done so in the previous 4 weeks;
6. Sunbed tanning or sunbathing in preceding 3 months, or planned sunbed tanning or sunbathing during the study period
7. Taking supplements known to have an effect on skin (e.g. fish oil, coenzyme Q-10, garlic, lycopene, beta-carotene, etc.), or have done so in the previous 4 weeks, except for medically-prescribed supplements or natural health products.
8. Supplements known not to have an effect on the skin (e.g. probiotics) are allowed, once the subject has been on a stable dose for greater than 3 months and are willing to continue this supplement for the duration of the study;
9. Systolic blood pressure ≥160 mmHg, diastolic blood pressure ≥100 mmHg. Subjects receiving blood pressure medications, must be on stable dose for greater than 3 months;
10. Known allergy to seafood;
11. Are hypersensitive to any of the components of the test product;
12. Disturbed absorption due to changes in the gastrointestinal tract (e.g., resections, diverticula, malabsorption, blind-loop syndrome);
13. Known alcohol abuse (> 21 units of alcohol per week) or drug abuse within the previous year of screening;
14. Clinically significant illness within 14 days prior to dosing;
15. Current or recent (within 3 months of screening visit) changes in diet, which in the opinion of the Investigator, deviates from a normal diet (e.g. vegetarians may be acceptable, vegans are not acceptable);
16. Planned major changes in life style (i.e. diet, dieting, exercise level, travelling) during the duration of the study;
17. Has any health conditions that would prevent from fulfilling the study requirements, put the subject at risk or would confound the interpretation of the study results as judged by the investigator on the basis of medical history and routine laboratory test results;
18. Are severely immunocompromised (HIV positive, transplant patient, on antirejection medications, on a steroid for >30 days, or chemotherapy or radiotherapy within the last year);
19. Experiences alarm features such as weight loss, rectal bleeding, recent change in bowel habit (<3 months) or abdominal pain;
20. Have a malignant disease or any concomitant end-stage organ disease;
21. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial;
22. Subjects receiving treatment involving experimental drugs. If the subject has been in a recent experimental trial, these must have been completed not less than 60 days prior to this study.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
To determine the effect of 12 weeks daily consumption of Superba Boost as compared to placebo on reduction in Trans-Epidermal Water-Loss (TEWL). | 12 weeks.
  Reduction in Trans-epidermal water loss (TEWL), measured at baseline and after 12 weeks of intervention using a TEWAMetre.

SECONDARY OUTCOMES:
To determine the effect of daily consumption of Superba Boost as compared to placebo on the reduction of Trans-epidermal water loss (TEWL), | 6 weeks.
  Changes in Trans-epidermal water loss (TEWL) from baseline to 6 weeks after start of treatment, using a TEWAMetre
To assess the effect of daily consumption of Superba Boost as compared to placebo on changes in skin hydration | 6 week
  Changes in skin hydration from baseline (pre-study) to 6 weeks after start of treatment using a Corneometer
To assess the effect of daily consumption of Superba Boost as compared to placebo on changes in skin hydration | 6 weeks
  Changes in skin hydration from 6 weeks of treatment until end-of-study using a Corneometer
To assess the effect of daily consumption of Superba Boost as compared to placebo on changes in skin firmness (6 weeks) | 6 weeks
  Changes in skin firmness from baseline (pre-study) to 6 weeks after start of treatment using a Cutometer
To assess the effect of daily consumption of Superba Boost as compared to placebo on changes in skin firmness | 6 weeks
  Changes in skin firmness from 6 weeks of treatment until end-of-study using a Cutometer
To assess the effect of daily consumption of Superba Boost as compared to placebo on changes on subjective evaluation | 6 weeks
  Subjective evaluation by study subjects, using questionnaires at 6 weeks of treatment
To assess the effect of daily consumption of Superba Boost as compared to placebo on changes on subjective evaluation | 12 weeks
  Subjective evaluation by study subjects, using visual analogue scale at 12 weeks of treatment lower scores indicating worse outcomes and higher scores indicating better outcomes.
To assess the effect of daily consumption of Superba Boost as compared to placebo on changes on Omega-3 index | 12 weeks
  Omega-3 index (%), using a blood spot collected by fingerpick

OTHER OUTCOMES:
To determine the effect of Superba Boost versus the placebo on the Lipid content of skin (Exploratory) | 12 weeks
  Skin content of the following lipids at week 6 and week 12 measured in pmol
  Analysis will be performed on the following lipids:
  * Nonhydroxydehydrosphingosine (NdS)
  * Nonhydroxysphingosine (NS)
  * Nonhydroxyphytosphingosine (NP)
  * Nonhydroxy-6-hydroxysphingosine (NH)
  * Alphahydroxydehydrosphingosine (AdS)
  * Alphahydroxysphingosine (AS)
  * Alphahydroxyphytosphingosine (AP)
  * Alphahydroxy-6-hydroxysphingosine (AH)
  * Omegahydroxysphingosine (EOS)
  * Omegahydroxyphytosphingosine (EOP)
  * Omegahydroxy-6-hydroxysphingosine (EOH)
  * Omegahydroxydehydrosphingosine (EOdS)
  * diacylglycerol
  * free cholesterol
  * cholesterol esters
  * triacylglycerols.

CONTACTS AND LOCATIONS:
Overall Officials: Sally O'Shea, MD, Principal Investigator — Atlantia Food Clinical Trials
Locations (1):
- Atlantia Food Clinical Trials, Cork, Munster, Ireland

IPD SHARING:
Plan to Share IPD: No